CLINICAL TRIAL: NCT01197014
Title: A Single-dose, Randomized, Two-period, Two-treatment, Two-sequence, Crossover Bioequivalence Study of Amlodipine and Losartan Versus Two Co-administration of Amlodipine and Losartan in Healthy Caucasian Subjects
Brief Title: A Bioequivalence Study of Amlodipine Plus Losartan Versus Amlodipine and Losartan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Kyung-mi Park / Director, Hanmi Pharmaceutical Company Limited.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10-ALOS-102
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Amlodipine, Losartan
MeSH Terms: interventions — Amlodipine; Losartan; amlodipine-losartan drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine plus Losartan (Experimental)
  Interventions: Drug: Amlodipine plus Losartan
- Amlodipine, Losartan (Active Comparator)
  Interventions: Drug: Amlodipine, Losartan

INTERVENTIONS:
Drug: Amlodipine plus Losartan — Amlodipine/Losartan high dose
  Arms: Amlodipine plus Losartan
Drug: Amlodipine, Losartan — Amlodipine, Losartan
  Arms: Amlodipine, Losartan

SUMMARY:
Study Design :

- A single center, open, randomized, single dose, two-period, two-treatment, two-sequence, crossover study

DETAILED DESCRIPTION:
Primary Objective:

- To assess the bioequivalence of combination oral formulation of amlodipine/losartan versus two co-administered products containing amlodipine and losartan

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Healthy Caucasian volunteers
* Non smokers or mild smokers

Exclusion criteria:

* Pregnancy and/or breast-feeding
* Participation in another clinical trial within 60 days prior to Period 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
AUC, Cmax | 0-144hrs

CONTACTS AND LOCATIONS:
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia